CLINICAL TRIAL: NCT02431481
Title: A Phase I, Open Label, Multicenter, Parallel-group, Single Dose Two-staged Study to Evaluate the Pharmacokinetics and Safety of a Single 400 mg Oral Dose of LEE011 in Subjects With Varying Degrees of Impaired Renal Function Compared to Matched Healthy Volunteers With Normal Renal Function
Brief Title: Evaluation of Renal Function Impairment on the Pharmacokinetics of LEE011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A2116
Record Dates: First submitted 2015-04-02; First posted 2015-05-01 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2019-02

CONDITIONS: Normal Renal Function; Impaired Renal Function
MeSH Terms: conditions — Renal Insufficiency | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Normal renal function (Experimental): Normal renal function; matched demography to renal impariment cohorts
  Interventions: Drug: LEE011
- Severe renal impairment (Experimental): Severe decrease in GFR (15-29 ml/min)
  Interventions: Drug: LEE011
- End Stage Renal Disease (Experimental): End stage renal disease not on dialysis; GFR <15 ml/min
  Interventions: Drug: LEE011
- Mild renal impairment (Experimental): Mild decrease in GFR (60-89 ml/min)
  Interventions: Drug: LEE011
- Moderate renal impairment (Experimental): Moderate decrease in GFR (30-59 ml/min)
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011 — 400 mg

SUMMARY:
The purpose of this study is to characterize the PK and safety profile of LEE011 following a single oral dose in adult subjects with various degrees of renal impairment compared to a matched group of healthy subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria (All Subjects):

* Male or female (sterile or postmenopausal) subjects between 18-75 (both inclusive) years of age and healthy as determined by absence of clinically significant deviation from normal in medical history, physical examination, vital signs, electrocardiograms, and clinical laboratory determinations (except for renal impaired subjects).
* Subjects must have a BMI between 18 kg/m2 and 38 kg/m2 and weight at least 50 kg and no more than 120 kg.
* Additional inclusion criteria for subjects with normal renal function:

  * An absolute GFR as determined by MDRD equation and conversion within normal range as determined by GFR > 90 mL/min

Inclusion Criteria (for subjects with impaired renal function):

- Subjects must have documented stable renal disease without evidence of renal progressive disease (stable renal disease is defined as no significant change, such as a stable absolute GFR, for 4 weeks prior to study entry.

Exclusion Criteria (All Subjects):

* Subject has received a renal transplant at any time in the past and is on immunosuppressant therapy
* History or presence of impaired cardiac function
* Any surgical or medical condition that may significantly alter the absorption, distribution, metabolism, or excretion of drugs
* Administration of CYP3A4/5 inhibitors or inducers or CYP3A4 substrates with narrow therapeutic windows
* Administration of medications that prolong the QT interval
* Subject has a history of immunodeficiency diseases, including HIV, as confirmed by (HIV-1, HIV-2) test
* Receipt of investigational product in another clinical trial within 4 weeks of dosing

Exclusion Criteria (for subjects with impaired renal function):

* Severe albuminuria > 300 mg/day
* Subjects undergoing any method of dialysis
* Subjects with renal impairment due to hepatic disease (hepatorenal syndrome)

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Primary Pharmacokinetics (PK) parameters of LEE011 when appropriate | 14 days
  Primary composite PK parameters: Cmax, AUClast, AUCinf, and CL/F. To determine the impact of various degrees of renal impairment on primary PK parameters of LEE011 following a single 400mg oral dose

SECONDARY OUTCOMES:
Secondary PK parameters of LEE011 when appropriate | 14 days
  Secondary composite PK parameters of LEE011: Tmax, T1/2, Vz/F, and CLr. To determine the impact of various degrees of renal impairment on secondary PK parameters of LEE011 following a single 400 mg oral dose
PK parameters of LEQ803 (i.e., Cmax, AUClast, AUCinf, Tmax, T1/2) | 14 days
  Composite PK parameters of LEQ803: Cmax, AUClast, AUCinf, Tmax, T1/2. To evaluate the PK profile of LEQ803 in subjects with various degrees of renal impairment following a single 400 mg oral dose
Frequency of adverse events (AEs) | From consent to 28 days post-dose
  Safety profile of a single dose of LEE011 in healthy subjects and subjects with varying degrees of hepatic function includes changes observed in physical examination, changes in vital signs, changes in electrocardiograms (ECGs), abnormal laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- DaVita Clinical Research, Minneapolis, Minnesota, United States
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Novartis Investigative Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111
- See also: Results for CLEE011A2116 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17418